CLINICAL TRIAL: NCT04986254
Title: A Multi-centre Study to Define Novel Individualised Dosing Regimens to Maximise Antibiotic Effectiveness for Treatment of Pneumonia in Intensive Care Units
Brief Title: PNEUmonia DOSing in Critically Ill Patients (PNEUDOS)
Acronym: PNEUDOS
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government); The Alfred (Other); University Hospital, Ghent (Other); Centre Hospitalier Universitaire de Nīmes (Other); Chinese University of Hong Kong (Other); University of Malaya (Other); International Islamic University Malaysia (Other); General Hospital of Larissa (Other); Central Hospital, Nancy, France (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PNEUDOS
Record Dates: First submitted 2021-07-06; First posted 2021-08-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia
Keywords: Pneumonia; Antibiotic dosing; Pharmacokinetic; Pharmacodynamic; Beta-lactam; Critically ill
MeSH Terms: conditions — Pneumonia; Critical Illness | interventions — Blood Specimen Collection; Ceftriaxone; Meropenem; Piperacillin; Tazobactam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each participant, samples of blood, epithelial lining fluid, and urine will be collected over 1 dosing interval (within the specified sampling times and time-points) on two separate occasions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Benzylpenicillin: ICU patients receiving benzylpenicillin for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically-diagnosed lung infection (n = 20)
  Interventions: Other: Blood sampling; Other: Epithelial lining fluid sampling; Other: Urine sampling; Drug: Study antibiotics include benzylpenicillin, ceftriaxone, meropenem, and piperacillin/tazobactam
- Ceftriaxone: ICU patients receiving ceftriaxone for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically-diagnosed lung infection (n = 20)
  Interventions: Other: Blood sampling; Other: Epithelial lining fluid sampling; Other: Urine sampling; Drug: Study antibiotics include benzylpenicillin, ceftriaxone, meropenem, and piperacillin/tazobactam
- Meropenem: ICU patients receiving meropenem for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically-diagnosed lung infection (n = 20)
  Interventions: Other: Blood sampling; Other: Epithelial lining fluid sampling; Other: Urine sampling; Drug: Study antibiotics include benzylpenicillin, ceftriaxone, meropenem, and piperacillin/tazobactam
- Piperacillin/tazobactam: ICU patients receiving piperacillin/tazobactam for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically-diagnosed lung infection (n = 20)
  Interventions: Other: Blood sampling; Other: Epithelial lining fluid sampling; Other: Urine sampling; Drug: Study antibiotics include benzylpenicillin, ceftriaxone, meropenem, and piperacillin/tazobactam

INTERVENTIONS:
Other: Blood sampling — During a single dosing interval, each participant will have 1 - 8 blood samples taken for each antibiotic. Blood samples (3 mL each) will be drawn from an existing arterial line or central venous catheter. Blood samples will be collected on 2 separate occasions; Occasion 1, between Days 1 - 3 of antibiotic therapy and Occasion 2, between Days 3 - 6 of antibiotic therapy.
Other: Epithelial lining fluid sampling — Epithelial lining fluid will be sampled using either a bronchoalveolar lavage (BAL) or mini-BAL technique, in accordance with the preferred procedure in participating sites. 3 BAL or mini-BAL samples will be collected over 2 separate occasions; Occasion 1, between Days 1 - 3 of antibiotic therapy and Occasion 2, between Days 3 - 6 of antibiotic therapy.
Other: Urine sampling — The total urine volume over the duration of the dosing interval will be collected on the two sampling occasions for a calculated urinary creatinine clearance measurement.
Drug: Study antibiotics include benzylpenicillin, ceftriaxone, meropenem, and piperacillin/tazobactam — Antibiotic dose and dosing interval will be determined by the treating clinician in accordance to standard prescribing practices based on clinical assessment of the patient. This study aims to recruit at least 20 participants per antibiotic.

SUMMARY:
Pneumonia is the most common infection in intensive care unit (ICU) patients and occurs in 10% of all ICU admissions. Unfortunately, ICU patient outcomes remain poor with a high mortality rate associated with pneumonia despite recent therapeutic advances.

Previous studies of antibiotics used in ICU patients, which includes ceftriaxone, meropenem and piperacillin/tazobactam, have quantified major differences in pharmacokinetics (PK) between ICU and non-ICU patients, with ICU patients displaying a unique spectrum of plasma concentration-time profiles. These PK differences can lead to suboptimal antibiotic concentrations in blood, which have been associated with a reduced likelihood of clinical cure for pneumonia. Furthermore, highlighting the importance of optimised dosing for pneumonia is that multi-drug resistant (MDR) pathogens emerge during antibiotic therapy in approximately half of the ICU patients, frequently emerging from the lung.

Previous work has highlighted how infection site concentrations determine patient outcome. For pneumonia, the infection site is best described as the epithelial lining fluid (ELF) in the lung.

Although optimal antibiotic therapy should be considered a priority for ICU patients with pneumonia to improve the persisting poor outcomes, the dosing regimens that can achieve therapeutic concentrations at the infection site (i.e., ELF) in ICU patients with pneumonia remain unknown.

The PNEUDOS study aims to address this significant knowledge gap by defining novel individualised dosing regimens that can maximise antibiotic efficacy by achieving therapeutic concentrations in the blood and ELF of ICU patients with pneumonia. These dosing regimens can then be validated in future clinical trials.

DETAILED DESCRIPTION:
Hypotheses

1. The pharmacokinetics of benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam are significantly different in ICU patients with pneumonia when compared to those of non-ICU and non-infected patients.
2. Altered beta-lactam antibiotic dosing approaches, as opposed to "contemporary" or "standard" dosing, are required for maximally effective blood (i.e., plasma) and epithelial lining fluid beta-lactam exposures in ICU patients with pneumonia.
3. Beta-lactam antibiotic exposures in epithelial lining fluid influence levels of lung inflammation in ICU patients with pneumonia.

Objective: The overall objective of this study is to characterise the plasma and epithelial lining fluid pharmacokinetics of important antibiotics in ICU patients with pneumonia to define optimal dosing regimens that maximise therapeutic outcomes.

Specific objectives

1. To describe the population pharmacokinetics of benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam (in plasma, epithelial lining fluid and urine) in ICU patients with pneumonia.
2. To design optimised dosing regimens for benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam that maximise the achievement of effective epithelial lining fluid exposures in ICU patients with pneumonia.
3. To characterise the effects of beta-lactam antibiotic (benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam) exposures in epithelial lining fluid on lung inflammation in ICU patients with pneumonia.

General design: This study is a prospective, open-labeled, multi-centre pharmacokinetic study, which is designed to develop an individualised and optimal dosing regimen for benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam in ICU patients with pneumonia.

Patient recruitment: An ICU patient who is receiving either benzylpenicillin, ceftriaxone, meropenem or piperacillin/tazobactam for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically diagnosed lung infection, who meets all the inclusion criteria and none of the exclusion criteria will be considered for study participation.

Study antibiotics

The study antibiotics include:

1. Benzylpenicillin
2. Ceftriaxone
3. Meropenem
4. Piperacillin/tazobactam

Antibiotic dose and dosing interval will be determined by the treating clinician in accordance to standard prescribing practices based on clinical assessment of the patient. This study aims to recruit at least 20 participants per antibiotic.

Study procedures: For each antibiotic, samples of blood, epithelial lining fluid and urine will be collected over one dosing interval (within the specified sampling times and time-points) on two separate occasions; Occasion 1, between Days 1 - 3 of antibiotic therapy and Occasion 2, between Days 3 - 6 of antibiotic therapy.

Blood sampling: During a single dosing interval, each participant will have 1 - 8 blood samples taken for each antibiotic. Blood samples (3 mL each) will be drawn from an existing arterial line or central venous catheter into heparinised tubes within the specified sampling times and time-points, in accordance with the method of antibiotic administration and dosing interval (i.e. intermittent infusion, extended infusion or continuous infusion).

Epithelial lining fluid sampling: Epithelial lining fluid will be sampled using either a bronchoalveolar lavage or mini-bronchoalveolar lavage technique, in accordance with the preferred procedure in participating sites. Where possible, epithelial lining fluid sampling will be performed on the same days and times as the blood sampling. Three bronchoalveolar lavage or mini-bronchoalveolar lavage samples will be collected over the two sampling occasions; Occasion 1, between Days 1 - 3 of antibiotic therapy and Occasion 2, between Days 3 - 6 of antibiotic therapy.

Urine sampling: The total urine volume over the duration of the dosing interval will be collected on the two sampling occasions for a calculated urinary creatinine clearance measurement.

Inflammatory cytokines/mediators in blood and epithelial lining fluid: Quantification of systemic and lung inflammation by measuring inflammatory cytokines/mediators such as C-reactive protein (CRP), interleukin-8 (IL-8), procalcitonin (PCT) and tumor necrosis factor-α (TNF-α) in blood and epithelial lining fluid will occur on sampling Occasion 1 and then again on Occasion 2. These samples will be used to determine CRP, IL-8, PCT and TNF-α, CRP and PCT levels.

Microbiological cultures: Bronchoalveolar lavage, blood or urine samples sent to the microbiology laboratory for culture as part of routine clinical care will be used to identify relevant causative organism(s) and drug susceptibility. Isolates of the identified causative organism will be transferred to the reference microbiological laboratory, University Queensland Centre for Clinical Research (UQCCR) at the University of Queensland so that the organism's minimum inhibitory concentration (MIC) can be determined using the broth microdilution and/or epsilometer test (Etest) methods, depending on clinical usage at the time of analysis.

Bioanalysis: Total and free drug concentrations in epithelial lining fluid, plasma and urine will be measured by a validated ultra-high performance liquid chromatography tandem mass spectrometry (UHPLC-MS/MS) method on a Nexera2 UHPLC system coupled to a 8050 triple quadruple mass spectrometer (Shimadzu Corporation, Kyoto, Japan). Bioanalysis will be conducted in accordance with U.S FDA guidance for industry on bioanalysis. Inflammatory cytokine/mediators will be measured by enzyme-linked immunosorbent assay (ELISA). Bioanalysis of samples will be conducted by Central Bioanalysis Laboratory at UQCCR, the University of Queensland.

Data collection: Data collection will be performed by trained personnel in the ICU and the data will be entered into an electronic case report form. The following parameters/variables will be collected from the patient medical record: (1) baseline variables; (2) ICU-related variables; (3) microbiological data; and (4) post-ICU variables (e.g. clinical cure on day of cessation of study antibiotic or at Day 14 post-enrolment).

Pharmacometric analysis plan Primary pharmacokinetic parameters (volume of distribution, Vd and clearance, CL) will be estimated. An attempt will be made to correlate any differences in these primary pharmacokinetics parameters between patients, with clinical and demographic characteristics of the patient. Variability in antibiotic dosing, infusion rates and sampling times will be accounted for by pharmacometric analyses and the software used to perform the analysis. Different dosing regimens, with various degrees of organ function and clinical characteristics, required to attain therapeutic concentrations at the site of infection will be evaluated using Monte Carlo dosing simulations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) ICU patients
2. Confirmed or suspected either community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically diagnosed lung infection
3. Patient has been prescribed or is receiving one of the study drugs (benzylpenicillin, ceftriaxone, meropenem, or piperacillin/tazobactam) for the treatment of pneumonia in the ICU
4. Patient is sedated and receiving mechanical ventilation
5. Patient has arterial line and urinary catheter in situ for blood and urine samplings
6. Informed consent to participate in the study

Exclusion Criteria:

1. Suspected or known hypersensitivity towards beta-lactam antibiotics (pre- or post-enrolment)
2. Receiving renal replacement therapy (RRT)
3. Pregnant patients or lactating mothers
4. Has received study antibiotic for more than 72 hours (at time of Occasion 1) during current infective episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A critically ill patient in the ICU who is receiving either benzylpenicillin, ceftriaxone, meropenem or piperacillin/tazobactam for confirmed/suspected community-acquired pneumonia, ventilator-associated pneumonia, aspiration pneumonia or a clinically diagnosed lung infection, who meets all the inclusion criteria and none of the exclusion criteria will be considered for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (Vd) of benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam in ICU patients with pneumonia | Days 1 - 6 of antibiotic therapy
  Population mean value of volume of distribution (Vd) in L/kg
Drug clearance (CL) of benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam in ICU patients with pneumonia | Days 1 - 6 of antibiotic therapy
  Population mean value of clearance (CL) in L/hr
Optimised dosing regimens for benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam that maximise the achievement of effective plasma exposure in ICU patients with pneumonia | Days 1 - 6 of antibiotic therapy
  Dosing regimens required to attain therapeutic concentrations in plasma will be evaluated using Monte Carlo dosing simulations. Therapeutic concentration is defined as concentrations above the minimum inhibitory concentration (MIC) of a pathogen for 100% of the dosing interval (100% T>MIC) in plasma
Optimised dosing regimens for benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam that maximise the achievement of effective epithelial lining fluid exposure in ICU patients with pneumonia | Days 1 - 6 of antibiotic therapy
  Dosing regimens required to attain therapeutic concentrations at the site of infection will be evaluated using Monte Carlo dosing simulations. Therapeutic concentration is defined as concentrations above the minimum inhibitory concentration (MIC) of a pathogen for 100% of the dosing interval (100% T>MIC) in the epithelial lining fluid
The effect of lung inflammation on beta-lactam antibiotic exposures | Days 1 - 6 of antibiotic therapy
  To characterise the effects of beta-lactam (benzylpenicillin, ceftriaxone, meropenem and piperacillin/tazobactam) exposures in epithelial lining fluid on lung inflammation (using inflammatory cytokines/mediators) in ICU patients with pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Jason A. Roberts, PhD, Principal Investigator — The University of Queensland
Locations (6):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane
  - The Alfred, Melbourne
- University Hospital, Ghent, Ghent, Belgium
- Centre Hospitalier Universitaire de Nimes, Nîmes, France
- Chinese University of Hong Kong, Hong Kong, Hong Kong
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdul-Aziz MH, Alffenaar JC, Bassetti M, Bracht H, Dimopoulos G, Marriott D, Neely MN, Paiva JA, Pea F, Sjovall F, Timsit JF, Udy AA, Wicha SG, Zeitlinger M, De Waele JJ, Roberts JA; Infection Section of European Society of Intensive Care Medicine (ESICM); Pharmacokinetic/pharmacodynamic and Critically Ill Patient Study Groups of European Society of Clinical Microbiology and Infectious Diseases (ESCMID); Infectious Diseases Group of International Association of Therapeutic Drug Monitoring and Clinical Toxicology (IATDMCT); Infections in the ICU and Sepsis Working Group of International Society of Antimicrobial Chemotherapy (ISAC). Antimicrobial therapeutic drug monitoring in critically ill adult patients: a Position Paper. Intensive Care Med. 2020 Jun;46(6):1127-1153. doi: 10.1007/s00134-020-06050-1. Epub 2020 May 7. PMID 32383061